CLINICAL TRIAL: NCT03556046
Title: An Open-label, Phase I Study to Assess Safety, Tolerability, Radiation Dosimetry, and Imaging Properties of 89Zr-labelled Girentuximab (89Zr-girentuximab) for in Vivo Detection of Clear Cell Renal Carcinoma (CCRC) by Positron Emission Tomography (PET) Using Different PET Imaging Methodologies
Brief Title: 89Zr-girentuximab ) Dosimetry in CCRC Study - ZIR-DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ABX CRO (Other); Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TLX-89Zr-TX-250-001D
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-05

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-girentuximab (Experimental): A single administration of 37 MBq (+/-10%) 89Zr-girentuximab, containing a mass dose of 5 mg of girentuximab
  Interventions: Diagnostic Test: 89Zr-Girentuximab

INTERVENTIONS:
Diagnostic Test: 89Zr-Girentuximab — Single diagnostic injection on Day 0, followed by diagnostic scans on Days 3 and 7±1, as well as the whole body dosimetric imaging on Days 0, 1, 3 and 7±1

SUMMARY:
The study is designed to explore the safety and tolerability as well as diagnostic 89Zr-girentuximab for imaging CCRC by PET/CT. This study does not offer any treatment for patients with CCRC; therefore, patients will be offered state of the art therapeutic options after imaging with the study drug 89Zr-girentuximab. Cancer treatment will not be delayed by study participation.

DETAILED DESCRIPTION:
The identification of RCC is crucial for planning possible surgery and treatment. The aim of this study is to investigate the safety, tolerability, radiation dosimetry, as well as the diagnostic performance of 89Zr-girentuximab PET/CT in patients with suspected CCRC. The results of this study will be used to pave the way for further studies with 89Zr-girentuximab as a PET/CT imaging agent which was shown to have higher diagnostic resolution 124I-girentuximab in animal studies due to prolonged trapping of the radiolabel in the tumour and simultaneous washout from normal tissues. It is anticipated to develop 89Zr-girentuximab as an improved imaging agent for CCRC.

This will be an exploratory, open-label, Phase 1 study to evaluate safety, tolerability, whole body dosimetry, and imaging properties of 89Zr-girentuximab, when image acquisition is made using different PET reconstruction methods, namely time-of-flight (TOF-PET) and conventional (PET) reconstruction, in order to estimate a possible impact of variable scanner technology on image quality variability in a planned multi-centre study.

In addition, different acquisition durations (5 -20 min) will be explored using an activity dose of 37 mBq (1 mCi), in order to establish, whether acquisition time has an impact on diagnostic performance.

It is anticipated to recruit 8-10 patients with suspected or established CCRC to

* Receive a slow intravenous injection with 89Zr-girentuximab (1-2 minutes slow bolus injection), followed by
* Dosimetric and tumour PET/CT imaging. The study duration will be approximately 12 months. Primary endpoint is safety, a part of which is determining the effective dose (mSv/MBq) to the whole body, and absorbed dose (mGy/MBq) to individually discernible organs.

Secondary endpoints include physicians assessment of PET image quality and tumour detectability comparing the following reconstruction settings:

TOF-PET PET 37 MBq 5, 10, 15 and 20 min 5, 10, 15 and 20 min Additionally, images partitioned to acquisition times of 5, 10, 15 and 20 min will be comparatively analysed in a blinded read.

In order to comprehensively characterise safety and tolerability, standard safety parameters (labs, 12-lead ECG, adverse events, and concomitant medications) will be systematically assessed at baseline and at appropriate intervals post dosing. Patients with clinical suspicion of CCRC, based on imaging evidence of a renal mass, requiring further diagnostic work-up, or patients with established diagnosis of CCRC requiring imaging for recurrent disease will be recruited by the urological service of the study centre, and undergo a formal screening visit, during which the study schedule will be planned, and consent obtained.

All successfully screened patients will be injected with 89Zr-girentuximab on Day 0 by the nuclear medicine service, followed by:

Sequential static whole body PET/CT imaging:

For dosimetry analysis, biodistribution whole body PET/CT imaging will be performed at 0.5, 4, 24, 72 and 168±24 h (Day 7±1) post injection, using low dose CT. Patients will be imaged on a TOF-PET scanner, offering the possibility of TOF (time-of-flight) and non-TOF reconstruction.

Comparative tumour PET/CT imaging:

On Days 3 and 7±1 (after the biodistribution whole body scans on Days 3 and 7), tumour imaging will be performed using gated or list mode acquisition, for generation of sub-partitioned data. Such data allow the mathematical generation of statistically independent images for various dose levels, based on the actual dose administered in the trial. Acquisition will be for 20 min.

An end of study visit will be conducted on Day 8±1. 89Zr-girentuximab dosimetry will be centrally analysed for absorbed organ and whole body doses in a standardised fashion. In addition, tumour absorbed doses will be determined for scientific purposes (estimation of achievable tumour doses of therapeutic nuclides labelled to girentuximab).

All image data analyses will be performed / confirmed centrally.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female >50 years of age
3. Clinical suspicion of CCRC, based on imaging evidence of a renal mass, requiring further diagnostic work-up or patients with established diagnosis of CCRC requiring imaging for recurrent disease
4. Life expectancy of at least 6 months
5. Consent to practise double-barrier contraception until end of study (7 days after 89Zr-girentuximab injection)

Exclusion Criteria:

1. Known hypersensitivity to girentuximab
2. Known uncontrolled hyperthyreoidism
3. Exposure to any experimental diagnostic or therapeutic drug within 30 days from the date of planned administration of 89Zr-girentuximab
4. Exposure to any radiopharmaceutical within 30 days (corresponding to 8 half-lives of 89Zr) prior to the administration of 89Zr-girentuximab.
5. Ongoing toxicity grade 2 from previous standard or investigational therapies (Common Terminology Criteria for Adverse Events [CTCAE] version 4.03)
6. Planned (for the period between injection of 89Zr-girentuximab and imaging) antineoplastic therapies
7. Established renal cell carcinomas of other histological entities than CCRC
8. Known brain metastases
9. Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic), that may interfere with the objectives of the study or with the safety or compliance of the patient, as judged by the investigator
10. Pregnant or breast-feeding women. Female patients of childbearing potential or male patients with female partners of childbearing potential, unless willing to practice full and true sexual abstinence or being surgically/permanently sterile or with a history of hysterectomy for women, not willing to practice effective double-barrier contraception by using: a non-oral, injected or implanted non-oestrogen progesterone based hormonal method, male condom, vaginal diaphragm, cervical cap, intrauterine device, during the study period and within a period of 30 days (corresponding to 8 half-lives of 89Zr) after receiving study drug.
11. Patients not able to declare meaningful informed consent on their own (e.g. with legal guardian for mental disorders)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Safety parameter Physical Examination | 8 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding the physical examination.
Safety parameter Vital Signs | 8 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding the Vital signs including the 12-lead ECG.
Safety parameter Adverse Events | 8 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding Adverse Events.
Safety parameter Laboratory examinations | 8 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding Laboratory examinations.
Safety parameter concomitant medications | 8 days
  Frequency of occurrence and severity of abnormal findings in safety investigations regarding concomitant medications.

SECONDARY OUTCOMES:
Radiation dosimetry | Whole body (neck to mid-thigh) static PET/CT scans will be acquired in supine position at 0.5, 4, 24, 72 and 168±24 h (Day 7±1) post injection, using low dose CT without contrast agent.
  Normalised whole body effective radiation dose (mSv/MBq)
Diagnostic efficacy | PET image acquisitions will be obtained in list mode on a TOF-capable machine for a period of 20 minutes.
  Visualisation of tumours will be qualitatively assessed across acquisition conditions (AC; i.e. reconstruction (Non-TOF/TOF), acquisition duration; details see above) by 2 readers experienced in oncology who will be blinded with regard to the AC.
  1. Percentage of images rated good or excellent / AC
  2. Percentage of images rated unevaluable / AC
  3. Total number of tumour lesions detectable / AC
  4. Comparative analysis of 5, 10, 15 and 20 min results at lesion basis.
Tumour dosimetry Absorbed dose | PET/CT, Days 3 (72 h) and 7(168 h)±1 post-infusion, with the contrast enhanced anatomical CT acquired as part of the baseline scan.
  Absorbed dose (Gy) from 89Zr-girentuximab to discernible tumour lesions, considering tumour volume, determined by pre-study contrast enhanced CT.
Tumour dosimetry Activity | PET/CT, Days 3 (72 h) and 7(168 h)±1 post-infusion, with the contrast enhanced anatomical CT acquired as part of the baseline scan.
  Determination of tumour tissue girentuximab exposure kinetics and AUC values (area under the curve), considering 89Zr-girentuximab specific activity at injection time point, injected activity, decay correction using the physical half-life of 89Zr, and anatomical tumour volume to obtain mg/mL.
Tumour dosimetry absorbed Dose | PET/CT, Days 3 (72 h) and 7(168 h)±1 post-infusion, with the contrast enhanced anatomical CT acquired as part of the baseline scan.
  Estimation of achievable absorbed tumour doses (Gy), assuming identical tumour biodistribution as observed for 89Zr-girentuximab, however therapeutic labelling with alpha and beta emitters.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tapner, Study Director — ABX CRO; Peter F. A. Mulders, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merkx RIJ, Lobeek D, Konijnenberg M, Jimenez-Franco LD, Kluge A, Oosterwijk E, Mulders PFA, Rijpkema M. Phase I study to assess safety, biodistribution and radiation dosimetry for 89Zr-girentuximab in patients with renal cell carcinoma. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3277-3285. doi: 10.1007/s00259-021-05271-w. Epub 2021 Mar 2. PMID 33651116